CLINICAL TRIAL: NCT02380352
Title: Short-course Antimicrobial Therapy for Paediatric Respiratory Infections
Acronym: SAFER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAFER 001 PSI; NCT01707485 (obsolete NCT alias)
Record Dates: First submitted 2015-03-02; First posted 2015-03-05 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Community-acquired Pneumonia
Keywords: antibiotic stewardship; non-inferiority; randomized controlled trial
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short-course (Experimental): 5 days amoxicillin 90 mg/kg/day divided TID followed by 5 days placebo TID
  Interventions: Drug: Amoxicillin; Drug: Placebo
- Standard (Active Comparator): 5 days amoxicillin 90 mg/kg/day divided TID followed by alternate formulation 5 days amoxicillin 90 mg/kg/day divided TID
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin
  Other Names: Amoxil
Drug: Placebo — Experimental arm must receive 5 days placebo after 5 days amoxicillin to preserve blinding.
  Arms: Short-course

SUMMARY:
Randomized controlled double-blind non-inferiority clinical trial to determine whether five days of high-dose amoxicillin leads to comparable rates of early clinical cure compared with 10 days of high-dose amoxicillin for previously healthy children with mild community-acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

Children aged 6 months to 10 years presenting with CAP will be eligible. CAP will be defined if all of the four following numeric criteria are met:

1. fever (>37.5 C axillary, > 37.7 C oral, or >38 C rectal) recorded in the ED or at home in the 48h prior to presentation;
2. any one of:

   1. tachypnoea on exam (>60 bpm for age <1 y, >50 bpm for 1-2 y of age, >40 bpm for 2-4 y of age, and >30 bpm for >4 y of age);
   2. cough on exam or by history;
   3. increased work of breathing on exam; or
   4. auscultatory findings (focal crackles, bronchial breathing, etc.) consistent with pneumonia;
3. infiltrates on chest radiograph consistent with bacterial CAP as judged by the ED physician; and
4. the attending ED physician diagnoses the child with primary CAP. (Children treated with systemic steroids in the ED will be presumed to have primary asthma exacerbation with possible infection and therefore will not meet inclusion criteria.)

Participants must be well enough to be treated as outpatients (discharged home by the ED physician, adequate volume status, able to tolerate oral medication, oxygen saturation > 90%, no evidence of impending respiratory failure), and have no evidence of empyaema or necrotizing pneumonia on chest radiograph.

Exclusion Criteria:

Children will be excluded if they have any of the following: cystic fibrosis, anatomic lung disease, bronchiectasis, congenital heart disease, history of repeated aspiration or velopharyngeal incompetence, malignancy, conditions requiring treatment with immune suppressants, primary immunodeficiency, advanced HIV infection, prolonged admissions (>48 h) to hospital within the past 2 months, pneumonia previously diagnosed within the past month, lung abscess diagnosed within the past six months, receipt of > 24 hours of beta-lactam antibiotic therapy already received at presentation to the ED, receipt of at least a 5 day course of amoxicillin < 72h prior to presenting to the ED, receipt of an intravenous cephalosporin or azithromycin in the ED, or suspected allergy to penicillin. Children will not be eligible to participate more than once.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 281 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Early clinical cure (Resolution of tachypnoea, increased work of breathing, and fever) | at 14-21 days post-enrolment
  Resolution of tachypnoea, increased work of breathing, and fever

SECONDARY OUTCOMES:
Days of adverse reactions | up to 14 days post-enrolment
Days of missed school | up to 14 days post-enrolment
Days of missed/disrupted work for caregiver(s) | up to 14 days post-enrolment
Adherence to study medications | up to 10 days post-enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Pernica, MD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario

REFERENCES:
- [Derived] Pernica JM, Harman S, Kam AJ, Carciumaru R, Vanniyasingam T, Crawford T, Dalgleish D, Khan S, Slinger RS, Fulford M, Main C, Smieja M, Thabane L, Loeb M. Short-Course Antimicrobial Therapy for Pediatric Community-Acquired Pneumonia: The SAFER Randomized Clinical Trial. JAMA Pediatr. 2021 May 1;175(5):475-482. doi: 10.1001/jamapediatrics.2020.6735. PMID 33683325
- [Derived] Pernica J, Harman S, Kam A, Bailey J, Carciumaru R, Khan S, Fulford M, Thabane L, Slinger R, Main C, Smieja M, Loeb M. Short-course antimicrobial therapy for paediatric respiratory infections (SAFER): study protocol for a randomized controlled trial. Trials. 2018 Feb 1;19(1):83. doi: 10.1186/s13063-018-2457-2. PMID 29391051